CLINICAL TRIAL: NCT02815644
Title: Investigation of the Effect of Food on the Bioavailability of Empagliflozin / Linagliptin Fixed Dose Combination Tablet in an Open, Randomised, Single Dose, Two Way Cross-over Study in Healthy Japanese Male Subjects
Brief Title: Empa/Lina FDC Food Effect Study (Japan)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1275.17
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Results first posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2017-10

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin

ARMS (1):
- empagliflozin/linagliptin FDC (Experimental): empagliflozin/linagliptin fixed-dose combination (FDC) film-coated tablet
  Interventions: Drug: empagliflozin/linagliptin FDC

INTERVENTIONS:
Drug: empagliflozin/linagliptin FDC — empagliflozin/linagliptin fixed-dose combination (FDC) film-coated tablet

SUMMARY:
The trial will be performed as an open-label, randomised, single-dose, two-sequence crossover design for the assessment of effect of food on bioavailability of empagliflozin / linagliptin fixed dose combination (FDC) tablet.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects age >=20 and <=45 years; body weight: >=50 kg and <=80 kg; body mass index: >=18.0 and <=25.0 kg/m2
* Without any clinically significant findings and complications on the basis of a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR), body temperature)
* Signed and dated written informed consent prior to admission to the trial in accordance with the Good Clinical Practice (GCP) and the local legislation

Exclusion criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and electrocardiogram) deviating from normal and of clinical relevance
* Further exclusion criteria apply

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2016-10-05 (Actual); Study Completion 2016-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a Open-label, randomised, single-dose, two-sequence, crossover design
Groups:
- Empagliflozin 25 mg/ Linagliptin 5 mg (Sequence 1: Fed-Fasted): Patient were orally administered Empagliflozin 25 mg/ linagliptin 5 mg fixed-dose combination (FDC) film coated tablet with 150 mL water after a standard Japanese breakfast in period 1 and after an overnight fast in period 2. Single-dose in each treatment period separated by wash-out period of at least 35 days
- Empagliflozin 25 mg/ Linagliptin 5 mg (Sequence 2: Fasted-Fed): Patient were orally administered Empagliflozin 25 mg/ linagliptin 5 mg fixed-dose combination (FDC) film-coated tablet with 150 mL water after an overnight fast in period 1 and after a standard Japanese breakfast in period 2. Single-dose in each treatment period separated by wash-out period of at least 35 days
Period: Treatment Period 1 + Washout
Arm/Group | Empagliflozin 25 mg/ Linagliptin 5 mg (Sequence 1: Fed-Fasted) | Empagliflozin 25 mg/ Linagliptin 5 mg (Sequence 2: Fasted-Fed)
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Empagliflozin 25 mg/ Linagliptin 5 mg (Sequence 1: Fed-Fasted) | Empagliflozin 25 mg/ Linagliptin 5 mg (Sequence 2: Fasted-Fed)
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This analysis set included all 22 randomised subjects who were documented to have taken at least 1 dose of trial medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin 25 mg/ Linagliptin 5 mg (Sequence 1: Fed-Fasted) | Empagliflozin 25 mg/ Linagliptin 5 mg (Sequence 2: Fasted-Fed) | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.00 (8.83) | 33.73 (9.55) | 31.36 (9.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Cmax for Linagliptin
Description: Maximum measured concentration of the analyte in plasma (Cmax) for linagliptin
Time Frame: 2 hours (h) before the administration in first subject and 0:20 h, 0:40h, 1:00h, 1:30h, 2:00h, 2:30h, 3:00h, 4:00h, 6:00h, 8:00h, 10:00h, 12:00h, 24:00h, 34:00h, 48:00h, 72:00h after drug administration.
Population: Pharmacokinetic Set (PKS): The PKS included all 22 randomised subjects who were documented to have taken at least 1 dose of trial medication under fed or fasted condition without having protocol deviation relevant to the evaluation of relative bioavailability and without experiencing emesis at or before 2 times median tmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- Empagliflozin 25 mg/ Linagliptin 5 mg (Reference;Fasted): Patient were orally administered Empagliflozin 25 mg/ linagliptin 5 mg fixed-dose combination (FDC) film coated tablet with 150 mL water after an overnight fast in period 1 or period 2. Single-dose in each treatment period separated by wash-out period of at least 35 days
- Empagliflozin 25 mg/ Linagliptin 5 mg (Test;Fed): Patient were orally administered Empagliflozin 25 mg/ linagliptin 5 mg fixed-dose combination (FDC) film-coated tablet with 150 mL water after a standard Japanese breakfast in period 1 or period 2. Single-dose in each treatment period separated by wash-out period of at least 35 days
Arm/Group | Empagliflozin 25 mg/ Linagliptin 5 mg (Reference;Fasted) | Empagliflozin 25 mg/ Linagliptin 5 mg (Test;Fed)
Number analyzed (Participants) | 22 | 22
nmol/L | 15.1 (50.6) | 8.43 (30.3)
Statistical Analysis 1: Comparison: Empagliflozin 25 mg/ Linagliptin 5 mg (Reference;Fasted) vs Empagliflozin 25 mg/ Linagliptin 5 mg (Test;Fed); Relative bioavailability of linagliptin after food intake compared to while in the fasting state was assessed using an ANOVA on the basis of the log transformed PK parameters. This model for the evaluation of effect of food on bioavailability included the effects: "sequence", "subjects within sequences", "period", and "treatment" (i.e., feeding status). The effect "subjects within sequences" was considered as random, whereas the other effects were considered as fixed; Test type: Superiority or Other; T/R ratio = 55.69, 90% CI 2-sided [48.22 to 64.33], Standard Error of Mean 1.087 — Standard Error of the mean is actually geometric Standard Error of the mean

2. Primary Outcome: Cmax for Empagliflozin
Description: Maximum measured concentration of the analyte in plasma (Cmax) for empagliflozin
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empagliflozin 25 mg/ Linagliptin 5 mg (Reference;Fasted) | Empagliflozin 25 mg/ Linagliptin 5 mg (Test;Fed)
Number analyzed (Participants) | 22 | 22
nmol/L | 1010 (27.1) | 756 (27.3)
Statistical Analysis 1: Comparison: Empagliflozin 25 mg/ Linagliptin 5 mg (Reference;Fasted) vs Empagliflozin 25 mg/ Linagliptin 5 mg (Test;Fed); Relative bioavailability of empagliflozin was assessed using an ANOVA on the basis of the log transformed PK parameters. This model for the evaluation of effect of food on bioavailability included the effects: "sequence", "subjects within sequences", "period", and "treatment" (i.e., feeding status). The effect "subjects within sequences" was considered as random, whereas the other effects were considered as fixed; Test type: Superiority or Other; T/R ratio = 74.89, 90% CI 2-sided [66.27 to 84.64], Standard Error of Mean 1.073 — Standard Error of the mean is actually geometric Standard Error of the mean

3. Primary Outcome: AUC 0-tz for Linagliptin
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable drug plasma concentration (AUC 0-tz) for linagliptin
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol∙h/L
Arm/Group | Empagliflozin 25 mg/ Linagliptin 5 mg (Reference;Fasted) | Empagliflozin 25 mg/ Linagliptin 5 mg (Test;Fed)
Number analyzed (Participants) | 22 | 22
nmol∙h/L | 348 (15.4) | 286 (20.5)
Statistical Analysis 1: Comparison: Empagliflozin 25 mg/ Linagliptin 5 mg (Reference;Fasted) vs Empagliflozin 25 mg/ Linagliptin 5 mg (Test;Fed); Relative bioavailability of linagliptin was assessed using an ANOVA on the basis of the log transformed PK parameters. This model for the evaluation of effect of food on bioavailability included the effects: "sequence", "subjects within sequences", "period", and "treatment" (i.e., feeding status). The effect "subjects within sequences" was considered as random, whereas the other effects were considered as fixed; Test type: Superiority or Other; T/R ratio = 82.19, 90% CI 2-sided [78.38 to 86.18], Standard Error of Mean 1.028 — Standard Error of the mean is actually geometric Standard Error of the mean

4. Primary Outcome: AUC 0-tz for Empagliflozin
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable drug plasma concentration (AUC 0-tz) for empagliflozin
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol∙h/L
Arm/Group | Empagliflozin 25 mg/ Linagliptin 5 mg (Reference;Fasted) | Empagliflozin 25 mg/ Linagliptin 5 mg (Test;Fed)
Number analyzed (Participants) | 22 | 22
nmol∙h/L | 7210 (19.1) | 6200 (20.6)
Statistical Analysis 1: Comparison: Empagliflozin 25 mg/ Linagliptin 5 mg (Reference;Fasted) vs Empagliflozin 25 mg/ Linagliptin 5 mg (Test;Fed); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; T/R ratio = 85.99, 90% CI 2-sided [83.38 to 88.68], Standard Error of Mean 1.018 — Standard Error of the mean is actually geometric Standard Error of the mean

5. Secondary Outcome: AUC0-infinity for Linagliptin
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-infinity) for linagliptin
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol∙h/L
Arm/Group | Empagliflozin 25 mg/ Linagliptin 5 mg (Reference;Fasted) | Empagliflozin 25 mg/ Linagliptin 5 mg (Test;Fed)
Number analyzed (Participants) | 22 | 22
nmol∙h/L | 597 (20.6) | 526 (33.4)
Statistical Analysis 1: Comparison: Empagliflozin 25 mg/ Linagliptin 5 mg (Reference;Fasted) vs Empagliflozin 25 mg/ Linagliptin 5 mg (Test;Fed); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; T/R ratio = 88.13, 90% CI 2-sided [80.89 to 96.03], Standard Error of Mean 1.051 — Standard Error of the mean is actually geometric Standard Error of the mean

6. Secondary Outcome: AUC0-infinity for Empagliflozin
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-infinity) for empagliflozin.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol∙h/L
Arm/Group | Empagliflozin 25 mg/ Linagliptin 5 mg (Reference;Fasted) | Empagliflozin 25 mg/ Linagliptin 5 mg (Test;Fed)
Number analyzed (Participants) | 22 | 22
nmol∙h/L | 7270 (19.1) | 6280 (20.4)
Statistical Analysis 1: Comparison: Empagliflozin 25 mg/ Linagliptin 5 mg (Reference;Fasted) vs Empagliflozin 25 mg/ Linagliptin 5 mg (Test;Fed); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; T/R ratio = 86.33, 90% CI 2-sided [83.61 to 89.13], Standard Error of Mean 1.019 — Standard Error of the mean is actually geometric Standard Error of the mean

7. Secondary Outcome: AUC0-72 for Linagliptin
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 72 hours (AUC0-72) for linagliptin
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol∙h/L
Arm/Group | Empagliflozin 25 mg/ Linagliptin 5 mg (Reference;Fasted) | Empagliflozin 25 mg/ Linagliptin 5 mg (Test;Fed)
Number analyzed (Participants) | 22 | 22
nmol∙h/L | 348 (15.4) | 286 (20.5)
Statistical Analysis 1: Comparison: Empagliflozin 25 mg/ Linagliptin 5 mg (Reference;Fasted) vs Empagliflozin 25 mg/ Linagliptin 5 mg (Test;Fed); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; T/R Ratio = 82.19, 90% CI 2-sided [78.38 to 86.18], Standard Error of Mean 1.028 — Standard Error of the mean is actually geometric Standard Error of the mean

ADVERSE EVENTS:
Time Frame: From first drug administration until 7 days thereafter for each treatment arm, up to 8 days
Arm/Group | Empagliflozin 25 mg/ Linagliptin 5 mg (Reference;Fasted) | Empagliflozin 25 mg/ Linagliptin 5 mg (Test;Fed)
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights